CLINICAL TRIAL: NCT03360617
Title: Safety Comparison of Antibiotics Administered Via Intravenous Push Versus Intravenous Piggyback to Adult Patients in the Emergency Department
Brief Title: Does a Safety Difference Exist Between IV Push and IV Piggyback Antibiotics?
Acronym: IVP-ABX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center of Southern Nevada (Other)
Responsible Party: Principal Investigator, Aryan Rahbar, PharmD, University Medical Center of Southern Nevada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UMC-2017-100
Record Dates: First submitted 2017-11-06; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Infection
Keywords: IV; Intravenous; IV Push; Piggyback; Antibiotics; Beta Lactam; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, double-blinded, double-dummy, randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: When the pharmacist prepares the medication he/she will refer to the randomization form to select the correct study arm. The pharmacist will place a protective cover over the syringe and over the piggyback bag before it is provided to the nurse administering the medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Syringe Arm (Experimental): IV antibiotics will be delivered by syringe IV push over 2-3 minutes
  Interventions: Device: Syringe IV Push over 2-3 minutes
- Piggyback Arm (Sham Comparator): IV antibiotics will be delivered by IV piggyback over 30 minutes
  Interventions: Device: Piggyback over 30 minutes

INTERVENTIONS:
Device: Syringe IV Push over 2-3 minutes — IV antibiotics will be administered by Syringe IV Push over 2-3 minutes
  Other Names: IVP
  Arms: Syringe Arm
Device: Piggyback over 30 minutes — IV antibiotics will be administered by IV Piggyback over 30 minutes.
  Arms: Piggyback Arm

SUMMARY:
This study compares whether or not a safety difference exists between delivering antibiotics via IV push or IV piggyback method.

DETAILED DESCRIPTION:
This study compares whether or not a safety difference exists between delivering antibiotics via the IV push or IV piggyback method. It will be a single center, prospective, double-blinded, double-dummy, randomized controlled trial on a convenience sample of patients presenting to the ED receiving select beta-lactam antibiotics. Patients will be randomized to IV push antibiotic plus IV piggyback placebo or IV push placebo plus IV piggyback antibiotic. Patients will only be enrolled when a pharmacist who is familiar with the study is available to prepare medications. Treatment group assignment will be predetermined using an Excel random number generator. An investigator will conduct an informed consent with the patient. Only the pharmacist will have access to the randomization records and will not reveal the randomization until the end of the study. If the patient consents to the study, a pharmacist involved in the study will prepare the IV push syringe and IV piggyback. The IV push syringe and IV piggyback will be prepared in a manner that makes the contents blinded. Preparation of the IV push syringe and IV piggyback are standardized. The syringe and piggyback will be handed to the nurse for administration. The IV push antibiotic will be administered over 2-3 minutes and the IV piggyback antibiotic will be administered over 30 minutes. The IV push and IV piggyback will be administered at the same time. A research assistant will conduct surveys with the patient at the start of administration and every 15 minutes for a total of 90 minutes to observe for any adverse drug reactions. During the 90-minute observation period, other medications will be allowed to be administered to the patient. All medications received during this time period will be documented in the patient data sheet. If an adverse drug reaction occurs, the attending physician or medical resident caring for the patient will be notified to come evaluate the patient. Adverse drug reaction severity will be determined by the attending physician or medical resident based on a predetermined scale. Adverse drug reaction information will be collected to determine correlation of adverse drug reaction to drug administration. Adverse drug reactions deemed as serious will be reported to the Institutional Review Board (IRB) within 5 days of the event.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patients who present to the adult ED in whom IV aztreonam, cefazolin, cefoxitin, ceftriaxone, cefepime, ertapenem, or meropenem is ordered by the treating physician

Exclusion Criteria:

* Pregnant or breastfeeding
* Non-English speaking patient
* Attending provider excludes patient
* Unable to consent
* Prisoner
* Allergy to any beta-lactam antibiotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Difference in number of adverse reactions at 90 minutes from time 0 | From the time of administration (time 0) to 90 minutes
  The difference in the number of adverse reactions between the study arms within the first 90 minutes following administration of antibiotics.

SECONDARY OUTCOMES:
Difference in severity of adverse reactions between study arms. | 90 minutes from drug administration (time 0)
  The difference in severity of adverse reaction between the study arms based on the National Cancer Institute's, Common Terminology Criteria for Adverse Events, v4.0 (2017)
Difference in adverse reaction type between study arms. | 90 minutes from drug administration (time 0)
  The difference between the study arms for type of adverse reactions based on the National Cancer Institute's, Common Terminology Criteria for Adverse Events, v4.0 (2017)
Difference in hospital length of stay between study arms | Time from subject's arrival to Emergency Department (ED) until either discharged from ED to home, or if admitted, hospital discharge up to 90 days from ED admission.
  The difference between the study arms hospital length of stay
Difference of In-Hospital Mortality between study arms | Time from the subject's arrival to the Emergency Department (ED) until the subject is pronounced dead up to 90 days from ED admission.
  The difference of in-hospital mortality between the study arms.
Cost comparison between study arms | 90 minutes from drug administration (time 0)
  A description of the cost of service between the study arms

CONTACTS AND LOCATIONS:
Overall Officials: Aryan Rahbar, PharmD, Principal Investigator — University Medical Center of Southern Nevada
Locations (1):
- University Medical Center of Southen Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garrelts JC, Wagner DJ. The pharmacokinetics, safety, and tolerance of cefepime administered as an intravenous bolus or as a rapid infusion. Ann Pharmacother. 1999 Dec;33(12):1258-61. doi: 10.1345/aph.19067. PMID 10630824
- [Background] Wiskirchen DE, Housman ST, Quintiliani R, Nicolau DP, Kuti JL. Comparative pharmacokinetics, pharmacodynamics, and tolerability of ertapenem 1 gram/day administered as a rapid 5-minute infusion versus the standard 30-minute infusion in healthy adult volunteers. Pharmacotherapy. 2013 Mar;33(3):266-74. doi: 10.1002/phar.1197. Epub 2013 Feb 11. PMID 23400916
- [Background] Poole SM, Nowobilski-Vasilios A, Free F. Intravenous push medications in the home. J Intraven Nurs. 1999 Jul-Aug;22(4):209-15. PMID 10476138
- [Background] Butterfield-Cowper JM, Burgner K. Effects of i.v. push administration on beta-lactam pharmacodynamics. Am J Health Syst Pharm. 2017 May 1;74(9):e170-e175. doi: 10.2146/ajhp150883. PMID 28438821
- [Background] Martz C, Hoesly M, Davis N. Reducing Order to Antibiotic Administration Time in Septic Patients: The Role of IV Push Antibiotics. Unpublished Abstract. Eastern Virginia Medical School Institutional Review Board.
- [Result] Institute for Safe Medication Practices (ISMP, 2015). Safe Practice guidelines for Adult IV Push Medications. Retrieved from http://www.ismp.org/Tools/guidelines/ivsummitpush/ivpushmedguidelines.pdf
- [Result] Rodriguez R. The Safety of Intravenous Drug Delivery Systems: Update on Current Issues Since the 2009 Consensus Development Conference. Hosp Pharm. 2018 Dec;53(6):408-414. doi: 10.1177/0018578718798638. Epub 2018 Sep 5. PMID 30559529
- [Result] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Crit Care Med. 2017 Mar;45(3):486-552. doi: 10.1097/CCM.0000000000002255. PMID 28098591
- [Result] Garrelts JC, Smith DF, Ast D, Peterie JD. A comparison of the safety, timing and cost-effectiveness of administering antibiotics by intravenous bolus (push) versus intravenous piggyback (slow infusion) in surgical prophylaxis. Pharmacoeconomics. 1992 Feb;1(2):116-23. doi: 10.2165/00019053-199201020-00008. PMID 10172048
- [Result] Norrby SR, Newell PA, Faulkner KL, Lesky W. Safety profile of meropenem: international clinical experience based on the first 3125 patients treated with meropenem. J Antimicrob Chemother. 1995 Jul;36 Suppl A:207-23. doi: 10.1093/jac/36.suppl_a.207. PMID 8543496